CLINICAL TRIAL: NCT01409681
Title: A Multi-Centered Trial Evaluating the Role of Vitamin D Metabolism in Non-Small Cell Lung Cancer
Acronym: EBUS
Status: Terminated | Type: Observational
Why Stopped: PI decided to terminate the study
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2010.105; HUM 44333 (Other: University of Michigan Health System IRB)
Record Dates: First submitted 2011-07-22; First posted 2011-08-04 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchial brush samples Bronchoscopy samples for RNA extraction and RT-PCR expression Blood samples
  * 7 mL for measurement of Serum total Vit-D levels and 1,25 (OH)2 D3 levels;
  * 5 ml collected in EDTA tube for CYP24A1 genotype analysis (common metabolizing agent for calcitriol) and CYP24 polymorphisms analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational Group: NSCLC subject undergoing bronchoscopy

SUMMARY:
Vitamin D exerts antiproliferative and differentiating effects in cancers, including non-small cell lung cancer (NSCLC). The active form of Vitamin D is 1,25, dihydroxycholecalciferol (calcitriol) which rapidly induces expression of cytochrome P450 24R-hydroxylase (CYP24A1). CYP24A1 initiates inactivation of calcitriol as a result of successive hydroxylation/oxidation reactions. This study seeks to prospectively determine the relationship between Vitamin D gene expression and median survival as a primary outcome, and between the Vitamin D receptor (VDR)/CYP24A1 gene expression and cancer stage, smoking status, serum 1,25 (OH)2D3 levels as well as CYP24A1 genotype.

DETAILED DESCRIPTION:
This study seeks to prospectively determine the relationship between Vitamin D gene expression and median survival as a primary outcome, and the relationships between the Vitamin D receptor (VDR)/CYP24A1 gene expression and cancer stage, smoking status, serum 1,25 (OH)2D3 levels as well as CYP24A1 genotype.

Patients who are suspected to have lung cancer will be recruited to this study prior to their diagnostic biopsy. Those who have consented to the study will give permission for blood and tissue from this biopsy to be analyzed for the study endpoints. Statistical analysis on this data will seek to correlate CYP24A1 expression and medican survival of the participants. Patients' data will be collected for smoking status and cancer stage.

Study enrollment to adequately power the study statistically is 80 patients. Anticipated study duration is from 12 months to 18 months for sample collection and two years for follow-up for patient survival.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for diagnostic bronchoscopy for suspected advanced stage lung cancer by CT/PET scanning.
2. Tumor or lymph node accessible by transbronchial needle aspiration.
3. Age 18-80.
4. All patients must be informed of the investigational nature of this study and must give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

1. Unstable cardiovascular disease or other systemic disease
2. Mental incompetence/active psychiatric illness
3. Medical contraindication for bronchoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early-stage non-small cell lung cancer undergoing a broncoscopy at the University of Michigan Health Center or at the Ann Arbor Veteran's Administration Hospital
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time to lung cancer related death | 18 months
  Time to lung cancer related death

CONTACTS AND LOCATIONS:
Overall Officials: Nithya Ramnath, MD, Principal Investigator — University of Michigan Medical Center and Veteran's Administration Health Center
Locations (2):
- United States (2):
  - United States Department of Veteran's Affairs Medical Center, Ann Arbor, Michigan
  - University of Michigan Cancer Center, Ann Arbor, Michigan